CLINICAL TRIAL: NCT03515421
Title: Project Frazier 3 Regulatory Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan Scotland Ltd (Industry)
Collaborators: Institute for Diabetes-Technology GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3165622
Record Dates: First submitted 2018-04-10; First posted 2018-05-03 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Glucose monitoring System (BGMS) (Experimental): Intervention: Blood Glucose monitoring Systems (BGMSs): Frazier 3 Verio and Frazier 3 UltraPLus.
  Results obtained from the BGMS for UP and SA are compared to a reference instrument (YSI)
  Interventions: Device: Frazier 3 Verio; Device: Frazier 3 UltraPlus

INTERVENTIONS:
Device: Frazier 3 Verio — In vitro diagnostic device (IVDD)
Device: Frazier 3 UltraPlus — In vitro diagnostic device (IVDD)

SUMMARY:
Clinical Evaluation of Blood Glucose Monitoring Systems (BGMSs)

DETAILED DESCRIPTION:
User performance, system use, system accuracy, user instruction for use and marketing claims evaluation of Blood Glucose Monitoring Systems.

ELIGIBILITY:
Summary of Inclusion Criteria

* Age - Subject is at least 12 years old.
* Informed Consent - Subject reads the appropriate Participant Information Sheet and signs the Informed Consent Form (section 12.0).
* Diabetes Diagnosis when applicable - type 1 or type 2 diabetes mellitus.
* Language - Subject reads and understands local language
* SMBG status confirmed
* Subject agrees to complete all aspects of the study

Summary of exclusion criteria

* Conflict of Interest
* Pregnancy - Subject is pregnant (as confirmed by Subject)
* User Performance Accuracy Testing - Technical Expertise

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
User Performance (UP) evaluation measured by blood glucose level (mg/dl) of BGMS vs reference instrument. | Up to 1 hour
  UP evaluation of blood glucose monitoring systems compared to a reference instrument. BGMSs samples collected by subject and reference samples collected by HCP ( Health Care Professional)
System Accuracy (SA) evaluation measured by blood glucose level(mg/dl) of BGMSs vs reference instrument. | Up to 1 hour
  Accuracy verification of blood glucose monitoring systems compared to a reference instrument. Samples collected by HCP only.
System Use Evaluation questionnaire | Up to 15 minutes
  Assessment of how the patient uses the BGMS.
Instructions for Use Evaluation questionnaire. | Up to 10 days.
  Questionnaires to assess the effectiveness of the instructions for use.
Marketing Claims Evaluation questionnaire. | Up to 10 days
  Assess Lay User Acceptance of the Frazier 3 BGMSs in support of marketing claims.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Stewart, Study Director — LifeScan Scotland
Locations (4):
- Institut für Diabetes-Technologie, Ulm, Germany
- United Kingdom (3):
  - Diabetes Centre, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Centre for Health Science, Inverness

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katz LB, Stewart L, Guthrie B, Cameron H. Patient Satisfaction With a New, High Accuracy Blood Glucose Meter That Provides Personalized Guidance, Insight, and Encouragement. J Diabetes Sci Technol. 2020 Mar;14(2):318-323. doi: 10.1177/1932296819867396. Epub 2019 Aug 2. PMID 31375031